CLINICAL TRIAL: NCT05882448
Title: Study of the Influence of Intraperitoneal Insufflation of Carbon Dioxide (CO2) by Laparoscopy on the Short-term Evolution of Premature Infants With Ulcerative Necrotizing Enterocolitis
Brief Title: Study of the Influence of Intraperitoneal Insufflation of CO2 by Laparoscopy on the Short-term Evolution of Premature Infants With Ulcerative Necrotizing Enterocolitis
Acronym: NECO2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP221170
Record Dates: First submitted 2023-04-24; First posted 2023-05-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Enterocolitis, Necrotizing
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Laparotomy; Laparoscopy

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: At the end of the operation, two dressings will be placed on the child's abdomen to ensure the blindness of the health professionals performing the postoperative care and the parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparotomy (Active Comparator): Exploratory and therapeutic laparotomy if necessary, in case of necrotic intestine requiring resection with anastomosis or stoma-type bowel diversion
  Interventions: Procedure: laparotomy
- Laparotomy and laparoscopy (Experimental): Exploratory and therapeutic laparotomy if necessary preceded by laparoscopy with insufflation of CO2 (placement of a 3mm trocar in the left hypochondrium and insufflation of a pneumoperitoneum (carbon dioxide, pressure: 6 mmHg, flow rate: 1.5 Liter/minute) for a duration of at least 5 minutes.
  Interventions: Procedure: laparotomy; Procedure: Laparoscopy

INTERVENTIONS:
Procedure: laparotomy — Exploratory and therapeutic laparotomy if necessary, in case of necrotic intestine requiring resection with anastomosis or stoma-type bowel diversion
Procedure: Laparoscopy — laparoscopy with insufflation of CO2 (placement of a 3mm trocar in the left hypochondrium and insufflation of a pneumoperitoneum (carbon dioxide, pressure: 6 mmHg, flow rate: 1.5 Liter/minute) for a duration of at least 5 minutes.
  Arms: Laparotomy and laparoscopy

SUMMARY:
Ulcerative-necrotizing enterocolitis (ECUN) is an infectious and inflammatory disease of the digestive tract, which can lead to intestinal necrosis or perforation.

This severe pathology of the newborn , often premature, requires urgent medical and surgical treatment in 25 to 50% of cases. The morbidity is high, both digestive and neurological. ECUN can lead to complications at short-term (death, intestinal stenosis) and at long-term (neuro-cognitive disorders). The challenge of preserving the neurological development is a major issue. It involves control of inflammation. This inflammation causes neurological lesions and is responsible for a disorder of the long-term neurocognitive development.

At Robert-Debré and Trousseau, the management of newborns with ECUN is focused on the control of this inflammation. A laparoscopy is performed first. The carbon dioxide (CO2) insufflated into the abdomen during a laparoscopy is thought to have an anti-inflammatory effect according to several experimental and clinical studies. A preliminary retrospective study at Robert-Debré showed a decrease in postoperative inflammation (decrease in C reactive protein at Day2 and Day 7 post-op) as well as a decrease in morbimortality (decrease in the rate of stoma and reoperation) in children who had a laparoscopic first operation compared to those who had a laparotomy alone. However, in many hospitals, laparotomy alone is currently the only surgical option.

This preliminary study may demonstrate that laparoscopy decreases early morbidity and mortality in children with ECUN through reduced inflammation, as reflected by postoperative C reactive protein.

DETAILED DESCRIPTION:
NECO2 is a pilot trial, evaluating the intermediate effectiveness to short/medium term of laparoscopy on the inflammatory reaction of premature newborns with complicated ECUN, requiring surgical treatment.

This is a multicenter randomized controlled trial in single blind, in two parallel arms, in ratio 1:1, of superiority.

This trial compares laparoscopy plus laparotomy versus laparotomy alone.

Children will be randomized into 2 groups:

* Laparoscopy + laparotomy group
* Laparotomy group

The main objective is to evaluate the inflammatory response Day 2 postoperative in preterm infants with ECUN who have undergone surgery.

The main criterion is the evolution of the blood C reactive protein level between Day 0 and Day 2 postoperatively.

The secondary objectives are:To evaluate in premature babies with ECUN who have had a surgical intervention (laparoscopy + laparotomy or laparotomy alone):

A.The postoperative biological inflammatory response at Day 7 B.Post-operative biological inflammatory response from Day 0 to Day 7 C.Post-operative mortality D.Post-operative bowel morbidity E.Post-operative re-intervention rate F.Length of hospital stay G.Post-operative neurological morbidity, medium term (corrected term 41 SA)

* To evaluate the tolerance of laparoscopy :

H.Intraoperative cardiorespiratory I.Loco-regional lesions linked to the insertion of the trocar

Secondary endpoints:

A. C reactive protein blood level at Day 7 B. Blood levels of Procalcitonin, Interleukin 6 and Tumor Necrosis Factor-alpha at Day 1, Day 2, Day 4, Day 7 C. Postoperative death from any cause D. Stoma rate, duration of parenteral nutrition, duration of hemodynamic support, duration of invasive ventilation (High frequency oscillatory ventilation/Synchronized Intermittent Mandatory Ventilation), Post-ECUN intestinal stenosis rate E. Re-intervention (laparotomy) and cause (post-ECUN stenosis, stoma closure) F. Length of hospital stay until return home G. Early postoperative neurological lesions observed on transfontanellar ultrasound and MRI at the corrected term of 41 weeks of amenorrhea, H. Oxygen saturation (SaO2), hypercapnia (pCO2) blood pressure (BP), cerebral oxygenation (Near InfraRed Spectroscopy (NIRS)) intraoperatively I. Intraoperative clinical monitoring: exploration of adjacent organs. Post-operative clinical monitoring: digestive signs monitoring of wounds until discharge.

Group 1: laparotomy only Group 2: laparotomy and laparoscopy

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn (term of birth: <37 weeks of amenorrhea)
* Diagnosis of ECUN by the surgeon (distension abdominal +/- rectal bleeding +/- green gastric residue, increased biological inflammatory syndrome, + pneumatosis on abdominal radiography)
* Hospitalized and complicated ECUN: presenting either a pneumoperitoneum on abdominal X-ray or a absence of clinical and biological improvement after 48 hours of maximum well-conducted medical treatment (IV antibiotic therapy and digestive rest).
* Hospitalized in the 2 participating centers
* Of which the 2 holders of parental authority have been informed and have signed the consent form
* Having social security coverage (social security or CMU)

Exclusion Criteria:

* Instability contraindicating movement to the operating room or contraindicating CO2 insufflation
* Diagnosis of isolated perforation of the small intestine (radiography:

pneumoperitoneum without pneumatosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
C reactive protein blood level | between Day 0 and Day 2 post surgery
  C reactive protein blood level

SECONDARY OUTCOMES:
Postoperative biological inflammatory reaction | Day 7 post surgery
  C reactive protein blood level
Specific post-operative biological inflammatory reaction | Day1, day 2, day 4 and day 7 post surgery
  Procalcitonin, Interleukin 6 and Tumor Necrosis Factor-alpha blood level
Postoperative mortality | up to 3 months
  Death due to any postoperative cause
Postoperative intestinal morbidity: stoma rate | up to 3 months
  Stoma rate
Postoperative intestinal morbidity: Duration of parenteral nutrition | up to 3 months
  Duration of parenteral nutrition
Postoperative intestinal morbidity: Duration of hemodynamic support | up to 3 months
  Duration of hemodynamic support
Postoperative intestinal morbidity: Duration of invasive ventilation (HFO: High frequency oscillatory ventilation/VACI: Synchronized Intermittent Mandatory Ventilation) | up to 3 months
  Duration of invasive ventilation (HFO: High frequency oscillatory ventilation/VACI: Synchronized Intermittent Mandatory Ventilation)
Postoperative intestinal morbidity: Rate of intestinal stenosis post-ECUN | up to 3 months
  Rate of intestinal stenosis post-ECUN
Postoperative reoperation rate | up to 3 months
  Reoperation (laparotomy) and cause (post ECUN stenosis, stoma closure)
Length of hospitalization | up to 3 months
  Duration of hospitalization until return home
Medium-term postoperative neurological morbidity | up to 3 months
  Early postoperative neurological lesions observed on transfontanellar ultrasound and MRI at term corrected for 41 weeks of amenorrhea
Oxygen saturation (SaO2) (Tolerance of laparoscopy (Intraoperative cardio-respiratory)) | During Surgery
  Oxygen saturation (SaO2)
Hypercapnia (pCO2) (Tolerance of laparoscopy (Intraoperative cardio-respiratory)) | During Surgery
  hypercapnia (pCO2)
Blood pressure (BP) (Tolerance of laparoscopy (Intraoperative cardio-respiratory)) | During Surgery
  blood pressure (systolic and diastolic)
Cerebral oxygenation (Near InfraRed Spectroscopy (NIRS)) (Tolerance of laparoscopy (Intraoperative cardio-respiratory)) | During Surgery
  cerebral oxygenation (Near InfraRed Spectroscopy (NIRS)) intraoperatively
Presence of loco-regional lesions related to the insertion of the trocar (Tolerance of laparoscopy) | up to 3 months
  Presence of loco-regional lesions related to the insertion of the trocar

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Armand Trousseau Service de Chirurgie Pédiatrique et Néonatale, Paris
  - Hôpital Robert Debré Service de Chirurgie Pédiatrique, Paris

IPD SHARING:
Plan to Share IPD: Undecided